CLINICAL TRIAL: NCT03645889
Title: Complementary Role of Herbal Traditional Chinese Medicine in Management of Mild to Moderate Childhood Asthma
Brief Title: Traditional Chinese Medicine in Management of Childhood Asthma
Acronym: TraCMAst
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: Singapore Thong Chai Medical Institution (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017/3129
Record Dates: First submitted 2017-12-28; First posted 2018-08-24 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2017-12

CONDITIONS: Asthma in Children
Keywords: Traditional Chinese Medicine
MeSH Terms: interventions — 1,2-dioleoyl-3-(9-(3-perylenoyl)nonanoyl)glycerol

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paediatric Lung Tonic (PLTG) (Experimental): Traditional Chinese Medicine (TCM) in granules dosage form to be dissolved for consumption.
  Interventions: Other: PLTG
- PLTG Placebo (Placebo Comparator): Starch granules with 10% TCM to mimic the colour, taste and smell of active TCM.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: PLTG — A combination of 13 herbal granules
  Arms: Paediatric Lung Tonic (PLTG)
Other: Placebo — 90% starch filler and 10% PLTG
  Arms: PLTG Placebo

SUMMARY:
Bronchial Asthma is a common childhood chronic disease characterized by chronic inflammation of the airways. Frequent relapse of asthma has serious impacts on the child's growth, impairs quality of life (QoL) and mortality, posing a huge economic burden on both family and society. According to Traditional Chinese Medicine (TCM) principles and theory, the main reason for children suffering from asthma are congenital deficiencies at birth which were not corrected and/or lack of appropriate care in the early childhood, leading to insufficiency of the lung, spleen and kidney, resulting in susceptibility to external pathogenic factors. During the interval phase of the illness, wheezing is not prominent and the "Lung-Spleen Qi Deficiency" (LSQD) syndrome is most commonly seen. TCM treatment aims to strengthen the body's immune system by nourishing the spleen, replenishing "Qi"(vital energy), tonifying the lungs and strengthening the exterior, thereby reducing incidences of relapse and improve QoL. It is hypothesized that TCM has adjuvant roles in the management of mild-moderate childhood asthma. Hence the primary aim of this study is to investigate the efficacy of using herbal TCM as adjuvant therapy in the management of symptoms and QoL in asthmatic patients. A randomized, double-blind cross-sectional, 2-arms placebo-controlled study will be carried out. Pediatric patients with mild-moderate asthma identified with LSQD will be randomized to either control or treatment group. Study participants in control group will continue their conventional western medicine (CWM) while those in TCM group will consume a decoction of herbal TCM for 12-weeks in addition to their CWM. Pulmonary function tests, Asthma Control Test, QoL and TCM questionnaires will be used as outcome measurement tools. In addition, liver and kidneys functions will be monitored for signs of toxicity.

DETAILED DESCRIPTION:
It is hypothesized that herbal Traditional Chinese Medicine (TCM) has adjuvant roles in the management of mild-moderate childhood asthma.

The primary aim of the study is to investigate the efficacy of using herbal TCM as adjuvant therapy in the management of symptoms and quality of life in asthmatic patients.

The secondary aim of the study is to investigate the improvement in pulmonary function test (PFT) and fractional exhaled nitric oxide (FeNO) test in asthmatic patients taking herbal TCM adjuvant therapy, and to monitor the safety profile of herbal TCM with regards to renal and liver functions.

ELIGIBILITY:
Inclusion Criteria:

* Have asthma which is partly controlled based on Global Initiative for Asthma (GINA) asthma control classification guideline and has Asthma Control Test (ACT) score ≥17 at point of recruitment.
* Currently using fluticasone as the only regular inhaled corticosteroid therapy for asthma control with fluticasone dosage ≤ 250mcg/day for at least past 3 months.
* Able to perform pulmonary function test
* Fulfil the TCM criteria of "lung-spleen qi deficiency " type of asthma

Exclusion Criteria:

* Laboratory results for renal and liver functions outside of normal range.
* Concomitant use of theophylline or montelukast.
* Concomitantly or in the last 3 months taking TCM
* Pregnant or lactation
* Known allergic reactions to food such as peanut, seafood, egg and milk

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Pediatric Asthma Quality of Life Change from Baseline at 3 months | 3 months
  Pediatric Asthma Quality of Life Questionnaire will be used to assess improvement in asthmatic symptoms and quality of life in patients receiving both conventional asthma treatment regimen and Traditional Chinese Medicine.

SECONDARY OUTCOMES:
Pulmonary Lung Function Change from Baseline at 3 months | 3 months
  Improvement in pulmonary lung function will be assessed using spirometry test.
Incidence of Treatment-Emergent Liver Associated Adverse Events | 3 months
  Clinical biochemistry tests to assess liver functions
Incidence of Treatment-Emergent Renal Associated Adverse Events | 3 months
  Clinical biochemistry tests to assess renal functions
Airway Inflammation Change from Baseline at 3 months | 3 months
  Reduction in factional exhaled nitric oxide as an indicator for improvement in airway inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Oon Hoe Teoh, MBBS, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No